CLINICAL TRIAL: NCT01868178
Title: Relationship Between Bispectral Index (BIS) and Spectral Entropy (SpEn) During Desflurane Anaesthesia
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Germano De Cosmo, PhD, Catholic University of the Sacred Heart
Other Study IDs: A 935/2007
Record Dates: First submitted 2012-11-12; First posted 2013-06-04 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-05

CONDITIONS: Intraoperative Awareness
Keywords: awareness
MeSH Terms: conditions — Intraoperative Awareness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- BIS Spectral Entropy Group: intraoperative monitoring with BIS and Spectral Entropy
  Interventions: Device: BIS and Spectral Entropy

INTERVENTIONS:
Device: BIS and Spectral Entropy — The aim of the study was investigated the effectiveness of Spectral Entropy and BIS in avoiding awareness

SUMMARY:
The aim of this study was to estimate the relationship between BIS and Spectral Entropy values and any explicit or implicit memory or dreams recall during desflurane anaesthesia.

DETAILED DESCRIPTION:
During the last decade, an increasing number of monitor systems were developed designed to assess the depth of anesthesia.

Awareness is a rare occurrence of explicit recalls during anaesthesia with an incidence of 0,18% and the use of cerebral monitoring prevents about 50% of these events.

Different stages of awareness should be defined and implicit memorization is subconscious awareness without explicit recall and possible implicit recall with an incidence greater than awareness.

To assess implicit recalls, a large number of test can be used, for example the "word stem completation test" and the "free recall association test". These result easy to use and reliable in detect implicit memory.

Bispectral Index (BIS) and Spectral Entropy (SpEn) has been proposed, in recent years, as electroencephalographic monitors of anaesthesia depth.

The bispectral index is a monitor of anaesthetic depth approved by the Food and Drug Administration in the USA. The BIS monitor reports a dimensionless number between 0 (complete EEG inactivity) and 100 (awake state); BIS values from 40 to 60 are thought to be suitable for general anaesthesia. Spectral Entropy acquires the electroencephalograph (EEG) and frontal electromyography (FEMG) signals which are processed into three parameters: State Entropy (SE), Response Entropy (RE) and Burst Suppression Ratio (BSR).

SE is computed over the EEG dominant part of the spectrum (0.8-32 Hz), and therefore primarily should reflect the cortical state of the patient and results useful to assess hypnotic effects of drugs .

RE is computed over a frequency range from 0.8 to47 Hz. It includes both the EEG-dominant and EMG-dominant part of the spectrum . The SE and RE values below 60 correlate with a low probability of consciousness. Also Bispectral Index provides BRS, an evaluation of burst suppression in which cerebral activity results suppressed.

BIS and Spectral Entropy are intended to decrease the risk of intraoperative awareness and to enable the anesthetist to reduce risk of the under- and overdosing of anesthetic agents and to ensure faster and more predictable wake-up and extubation.

Previous studies result contrasting in the correlation between these devices with lack in evaluation of implicit memory.

The aim of this study was to estimate the relationship between BIS and Spectral Entropy values and any explicit or implicit memory or dreams recall during desflurane anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologist physical status I-II
* Italian native speakers

Exclusion Criteria:

* Psychiatric or neurologic diseases
* Acoustic impairment
* Obesity (Body Mass Index > 30)
* Substance dependence.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: female patients, aged 30-60 years , scheduled for minor elective surgery lasts between 1 and 3 hours were enrolled.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
BIS index | change from baseline at 15 min

SECONDARY OUTCOMES:
entropy values | 24 h after emergency from anaesthesia

OTHER OUTCOMES:
explicit and implicit memory and dreams recall. | after 24 h

CONTACTS AND LOCATIONS:
Overall Officials: De Cosmo Germano, PhD, Principal Investigator — Catholic University of Sacred Heart
Locations (2):
- Italy (2):
  - Catholic University of Sacred Heart, Rome, Rm
  - Catholic University, Rome, Rm

REFERENCES:
- [Background] Domino KB, Posner KL, Caplan RA, Cheney FW. Awareness during anesthesia: a closed claims analysis. Anesthesiology. 1999 Apr;90(4):1053-61. doi: 10.1097/00000542-199904000-00019. PMID 10201677
- [Background] Heier T, Steen PA. Awareness in anaesthesia: incidence, consequences and prevention. Acta Anaesthesiol Scand. 1996 Oct;40(9):1073-86. doi: 10.1111/j.1399-6576.1996.tb05569.x. PMID 8933848
- [Background] Liu WH, Thorp TA, Graham SG, Aitkenhead AR. Incidence of awareness with recall during general anaesthesia. Anaesthesia. 1991 Jun;46(6):435-7. doi: 10.1111/j.1365-2044.1991.tb11677.x. PMID 2048657
- [Background] O'Connor MF, Daves SM, Tung A, Cook RI, Thisted R, Apfelbaum J. BIS monitoring to prevent awareness during general anesthesia. Anesthesiology. 2001 Mar;94(3):520-2. doi: 10.1097/00000542-200103000-00025. PMID 11374615
- [Background] Brice DD, Hetherington RR, Utting JE. A simple study of awareness and dreaming during anaesthesia. Br J Anaesth. 1970 Jun;42(6):535-42. doi: 10.1093/bja/42.6.535. No abstract available. PMID 5423844
- [Background] Ranta SO, Laurila R, Saario J, Ali-Melkkila T, Hynynen M. Awareness with recall during general anesthesia: incidence and risk factors. Anesth Analg. 1998 May;86(5):1084-9. doi: 10.1097/00000539-199805000-00035. PMID 9585303
- [Background] Ghoneim MM. Incidence of and risk factors for awareness during anaesthesia. Best Pract Res Clin Anaesthesiol. 2007 Sep;21(3):327-43. doi: 10.1016/j.bpa.2007.05.002. PMID 17900012
- [Background] Kissin I. Depth of anesthesia and bispectral index monitoring. Anesth Analg. 2000 May;90(5):1114-7. doi: 10.1097/00000539-200005000-00021. No abstract available. PMID 10781463
- [Background] Paolo Martorano P, Falzetti G, Pelaia P. Bispectral index and spectral entropy in neuroanesthesia. J Neurosurg Anesthesiol. 2006 Jul;18(3):205-10. doi: 10.1097/01.ana.0000206229.38883.d2. PMID 16799349
- [Background] Liu J, Singh H, White PF. Electroencephalographic bispectral index correlates with intraoperative recall and depth of propofol-induced sedation. Anesth Analg. 1997 Jan;84(1):185-9. doi: 10.1097/00000539-199701000-00033. PMID 8989022